CLINICAL TRIAL: NCT00628849
Title: A Comparison of 2mm Plates and Screws With Larger Plates Ans Screws in the Treatment of Mandibular Fractures
Brief Title: Champy Versus AO for Mandible Fractures
Acronym: Mand
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Gary F Bouloux MD, DDS, MDSc, FRACDS, FRACDS, Principal Investigator, Emory University
Other Study IDs: IRB00000444
Record Dates: First submitted 2008-02-15; First posted 2008-03-05 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Mandibular Injuries
Keywords: Mandible; fracture; Champy; AO technique
MeSH Terms: conditions — Mandibular Injuries; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: This group will have 2 mm plates and screws placed according to Champy principles
- 2: This group will have 2 mm plates placed according to modified Champy principles
- 3: This group will have larger (2.3 mm or greater) plates and screws placed according to the AO technique

SUMMARY:
Patients who sustain a broken lower jaw have traditionally been treated in one of three ways. The first involves having their teeth and jaws being wired together for a period of 4 to 6 weeks in order to allow the broken jaw to heal. The second and third ways involve a surgical procedure that requires exposing the broken bones and stabilizing them with metal plates and screws that allow the patient to be able to function relatively normally during the healing period. One surgical method uses small plates and screws while the alternate method uses large plates and screws. Currently there are two schools of thought with respect to what plates and screws should be used. One group supports the use of large rigid plates due to the increased strength of the plate. The use of the larger and stronger plates is the principle behind the AO technique, which was originally developed in the 1970's in Switzerland and is now the more popular technique in the USA. The other group supports the use of smaller plates and screws which must be placed in certain anatomical positions to allow the natural muscular forces that exist on the jaw to stabilize the break and facilitate complete healing of the broken bone. This technique was developed in France by Maxime Champy in the 1970's and is the standard of care throughout Australasia and parts of Europe. This technique is simpler, quicker and cheaper. The need for patients to maintain a diet with softer foods is considered by many to be important for success if the less rigid and smaller plates are going to be used. Many critics of the Champy technique feel that less compliant patient populations as might be seen in a county hospital make the technique less readily suited to these populations. This is contrary to published data from Europe, Australia and recently the USA.

The question of interest is whether the smaller plates and screws are equally as effective in the treatment of broken lower jaws in an urban county hospital? If they are equally effective, then is there any benefit in terms of fewer patient complications and decreased health costs? If the smaller plates and screws are not adequate, then will a modification of the original Champy technique improve their usefulness? Patients who present with a broken lower jaw who require surgery will be treated in one of three ways. Some patients will be treated with the larger plates and screws by an attending surgeon who routinely uses large plates and screws for broken lower jaws. Another group of patients will be treated with the smaller plates and screws using the Champy principles. A third group of patients will also be treated with the smaller plates and screws but using a modification of the original Champy technique that involves the use of additional small plates and screws for added stability. Patients will then be followed over a three month period to evaluate for healing of the broken jaw. The three techniques will be then be compared.

Larger plates/ screws and the smaller plates/ screws are both the standard of care. Regional differences throughout the USA has continued to ensure differences of opinion with regard to which technique is better although historically the larger plates/screws has been more popular in the USA.

DETAILED DESCRIPTION:
All patients will have ORIF of their fractured mandible under general anesthesia. Patients will either be treated with small 2 mm plates and screws according to Champy principles (or a modified Champy technique that utilizes additional 2mm plates/screws) or larger plates/screws (2.3mm or larger) according to the AO principles. No patients will have their teeth wired together so that all patients will be able to function normally. All patients will have an immediate post operative orthopantogram to verify adequacy of the fracture reduction. Patients will be discharged as soon as is medically appropriate.

Patient Assessment

Patients will be assessed regularly at 1 week, 3 weeks, 6 weeks and 3 months to ensure continued healing of the fracture. This is a typical post-operative follow-up schedule for all fracture patients. As is the standard of care, orthopantogram x-rays will be taken at 6 weeks and 3 months to assess fracture healing. Additional x-rays will only be taken if the clinical picture is suggestive of inadequate healing or infection. Additional data regarding the presence of infection, nonunion, fibrous union, malunion, malocclusion, facial nerve weakness and inferior alveolar nerve paresthesia will be recorded at each follow-up visit. Additional complications will also be recorded and managed as necessary.

ELIGIBILITY:
Inclusion Criteria:

* all patients with a fractured mandible
* age 11 to 89

Exclusion Criteria:

* Comminuted fractures

Ages: 11 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who present with a fractured mandible
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2007-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
fracture healing | 3 months

SECONDARY OUTCOMES:
malocclusion | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gary F Bouloux, MD, DDS, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States